CLINICAL TRIAL: NCT04576910
Title: Immunogenicity and Safety of the Booster Dose of Polio Vaccine Immunization Using Sabin IPV or bOPV at Children Aged 4 Years With Different Three Sequential Schedules History by Sabin IPV or bOPV in China
Brief Title: Immunogenicity and Safety of the Booster Dose of Polio Vaccine With Different Primary Sequential Schedules in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Collaborators: China National Biotec Group Company ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZJCDC202002701
Record Dates: First submitted 2020-09-18; First posted 2020-10-06 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Polio; Vaccine Reaction
Keywords: Immunogenicity; Antibody persistence; Safety; Sabin IPV; bOPV
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A("Sabin IPV+ bOPV+ bOPV"+Sabin IPV) (Experimental): Give the 4th doses of polio vaccine with Sabin IPV for participants in the Group 1 of preliminary study (NCT03147560).
  Interventions: Biological: vaccinated with Sabin IPV
- Group B("Sabin IPV+ Sabin IPV+ bOPV"+bOPV) (Experimental): Give the 4th doses of polio vaccine with bOPV for participants in the Group 2 of preliminary study (NCT03147560) after randomization.
  Interventions: Biological: vaccinated with bOPV
- Group C("Sabin IPV+ Sabin IPV+ bOPV"+Sabin IPV) (Experimental): Give the 4th doses of polio vaccine with Sabin IPV for participants in the Group 2 of preliminary study (NCT03147560) after randomization.
  Interventions: Biological: vaccinated with Sabin IPV
- Group D("Sabin IPV+ Sabin IPV+ Sabin IPV"+bOPV) (Experimental): Give the 4th doses of polio vaccine with bOPV for participants in the Group 3 of preliminary study (NCT03147560) after randomization.
  Interventions: Biological: vaccinated with bOPV
- Group E("Sabin IPV+ Sabin IPV+ Sabin IPV"+Sabin IPV) (Experimental): Give the 4th doses of polio vaccine with Sabin IPV for participants in the Group 3 of preliminary study (NCT03147560) after randomization.
  Interventions: Biological: vaccinated with Sabin IPV

INTERVENTIONS:
Biological: vaccinated with Sabin IPV — the 4th dose of polio vaccination
  Arms: Group A("Sabin IPV+ bOPV+ bOPV"+Sabin IPV); Group C("Sabin IPV+ Sabin IPV+ bOPV"+Sabin IPV); Group E("Sabin IPV+ Sabin IPV+ Sabin IPV"+Sabin IPV)
Biological: vaccinated with bOPV — the 4th dose of polio vaccination
  Arms: Group B("Sabin IPV+ Sabin IPV+ bOPV"+bOPV); Group D("Sabin IPV+ Sabin IPV+ Sabin IPV"+bOPV)

SUMMARY:
This study is to evaluate the immunogenicity and safety of Sabin IPV or bOPV, given as a booster vaccination in children aged 4 years who were previously immunised with different sequential immunization history by Sabin IPV and bOPV, and to observe the antibody persistence three years after different primary sequential immunization with Sabin IPV or bOPV at age 2, 3 and 4 months.

DETAILED DESCRIPTION:
This is a continuous study of preliminary trial (Immunogenicity of three sequential schedules with Sabin inactivated poliovirus vaccine and bivalent oral poliovirus vaccine in Zhejiang, China: NCT03147560) . The investigators will follow up previous participants at age 4 years old with different primary sequential immunization schedules at age 2, 3 and 4 months: sIPV-bOPV-bOPV , sIPV-sIPV-bOPV , or sIPV-sIPV-sIPV, and give the 4th doses of polio vaccine with Sabin IPV or bOPV. A pre-vaccination blood sample is taken for polio antibody determinations. Sabin IPV will be administrated for participants in the previous Group 1 (sIPV-bOPV-bOPV), and Sabin IPV or bOPV will be given for participants in the previous Group 2 (sIPV-sIPV-bOPV) and Group 3 (sIPV-sIPV-sIPV) after they were randomly divided into two subgroups. At least two active surveillance visits, during which staff visited the participants s at home (on days 3 and 30) will required after vaccination to collect adverse reaction data. Parents or legal guardians were instructed to contact investigators if they observed any possible vaccine-related adverse events or important medical events (such as serious illness, physical disability, or death). The second blood sample will be collected 28-60 days after the booster vaccination. The investigators will asess the immunogenicity by seroconversion rate and seropositivity after the booster vaccination, and evaluate the antibody persistence using seropositive rate and GMT in participants before the booster vaccination. Safety will assessed with the occurrence of adverse events reported across the study groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥48 months to ≤ 51 months from preliminary study (NCT03147560) with sequential immunization history by Sabin IPV and bOPV.
* Parent/legal acceptable representative is willing and able to understand the protocol requirements and provide informed consent.
* ≥ 14 days interval between the last vaccination.
* Body temperature ≤ 37.2℃.

Exclusion Criteria:

* Known acute illness, severe chronic disease, acute exacerbation of chronic disease and fever.
* Known allergy to any constituent of the vaccine.
* Had 4 doses vaccination record of polio vaccine.
* Known impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin .
* Received non-specific immunoglobulin within 1 month.
* An acute illness with fever (temperature ≥ 37.3℃) or any infectious diseases.
* Patients with a well-diagnosed history of thrombocytopenia or other coagulation disorders that may cause contraindications for injection.
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the vaccine.

Ages: 48 Months to 51 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 387 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates of the booster vaccination | before and 28-60 days after the booster dose (4 years old) of polio vaccine
  Defined as any positive antibody (titre ≥ 8) response in children who were seronegative prior to the vaccination, or at least a fourfold increase in type-specific antibody levels for children who had pre-existing positive antibodies
Persistence (tite rates) of antibodies against poliovirus 3 years after the primary 3 dose polio vaccine immunization | 3 years after the primary three doses of polio immunization(before the booster vaccination )
  The percentage of participants with positive antibody(titre ≥ 8) against all three serotypes of poliovirus 3 years after the primary immunization with different sequential immunization schedules using sIPV or bOPV
Seroprotection rates after the booster vaccination | 28-60 days after the booster dose (4 years old) of polio vaccine
  The percentage of participants with positive antibody(titre ≥ 8) against all three serotypes of poliovirus

SECONDARY OUTCOMES:
Safety of the booster dose of polio vaccine immunization | 30 days after the booster vaccination
  the occurrence of adverse events for the booster dose of Polio vaccine administered at age 4 using Sabin IPV or bOPV
Antibody titers pesistence against poliovirus | 3 years after the primary three doses of polio immunization(before the booster vaccination )
  Geometric Mean Titres (GMTs) or Median antibody titers for three poliovirus types
Antibody titers against poliovirus after the booster immunization | 28-60 days after the booster dose of polio vaccine given
  Geometric Mean Titres (GMTs) or Median antibody titers for three poliovirus types after the booster dose of Polio vaccine administered at age 4 using Sabin IPV or bOPV

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chunan center for disease control and prevention, Hangzhou, Zhejiang
  - Longyou Center for Disease Control and Prevention, Quzhou, Zhejiang

REFERENCES:
- [Derived] Tang X, Xiao Y, Deng X, Zhou Y, Chen H, Yan R, Zhu Y, Wang S, Wang H, Zhu X, Luo L, Liu Y, Yin Z, Zhang G, Chen Z, Jiang J, Yang X, He H. Immuno-persistence of the different primary polio vaccine schedules and immunogenicity of the booster dose by sabin inactivated or bivalent oral poliovirus vaccine in children aged 4 years: an open-label, randomised, controlled phase 4 trial in China. Lancet Reg Health West Pac. 2023 Mar 17;34:100725. doi: 10.1016/j.lanwpc.2023.100725. eCollection 2023 May. PMID 37283972